CLINICAL TRIAL: NCT03202693
Title: A Phase 1, Open-Label, Single-Dose Study of the Safety, Tolerability, and Absorption, Metabolism, and Excretion of [14C]-PA 824 in Healthy Adult Male Subjects.
Brief Title: A Study of the Safety, Tolerability, and Absorption, Metabolism, and Excretion of PA-824 in Healthy Adult Male Subjects.
Acronym: CL-004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA 824-CL-004
Record Dates: First submitted 2017-06-01; First posted 2017-06-28 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, PA-824
MeSH Terms: conditions — Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PA-824 (Experimental): [14C]-PA-824 and unlabelled PA-824 oral suspension of 1000 mg unlabeled micronized PA-824 mixed with sufficient [14C]-PA-824 to achieve a final radiolabel dose of approximately 100 µCi/dose.
  Interventions: Drug: PA-824

INTERVENTIONS:
Drug: PA-824

SUMMARY:
This study is a Phase 1, single-center, open-label, single-dose study to evaluate (1) the absorption, metabolism, and excretion patterns of a single dose of [14C] PA-824, and (2) the pharmacokinetics, safety, and tolerability of a single oral-suspension dose of unlabeled PA-824 in healthy adult male subjects. Unlabeled PA-824 and [14C]-PA-824 will be administered together in an oral-suspension formulation. Enrollment is planned for one dose group of 6 subjects. All 6 subjects will receive the same treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be healthy non-tobacco/nicotine using (6-month minimum) adult male subjects, 19 to 50 years of age, inclusive
2. Weigh within 20% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1999)
3. Be medically healthy subjects with clinically insignificant Screening results (among laboratory profiles, medical histories, ECGs, or physical exam), as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
4. Have a history of regular bowel movements (5-6 movements week, ideally 1 per day), as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
5. Have negative urinalysis test results for drugs of abuse such as amphetamines, cannabinoids, and cocaine metabolites
6. Have the ability to understand the requirements of the study, have provided written informed consent (as evidenced by signature on an informed consent document approved by an IRB), and agree to abide by the study restrictions

Exclusion Criteria:

1. Any acute illness or history or presence of significant (as deemed by the Principal Investigator) cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
2. Any preexisting condition that would interfere with normal anatomy or function of the gastrointestinal tract.
3. Any medical condition that would interfere with radiocarbon assessments.
4. Any serum creatinine or BUN measure beyond the upper limit of the normal range at Screening or Check-in.
5. Positive Screening test for HCV, HBV, or HIV
6. History of peptic ulcer disease, gastritis, esophagitis, or gastroesophageal reflux disease
7. History of any cardiac abnormality (as deemed by the Principal Investigator)
8. History of hypokalemia or hypomagnesemia
9. History of prolonged QT interval
10. Family history of Long-QT Syndrome or sudden death
11. Resting pulse rate < 40 or > 100 bpm at both Screening and Check-in
12. QTc interval > 430 msec as documented at Screening and Baseline (Check-in) ECG
13. History or presence of alcoholism or drug abuse within the past year (as deemed by the Principal Investigator)
14. Use of alcohol within 72 hours prior to dosing
15. Significant history of drug and/or food allergies (as deemed by the Principal Investigator)
16. Use of any prescription medication within 14 days prior to dosing or during the study
17. Use of any over-the-counter medication including vitamins, herbal preparations, antacids, cough and cold remedies, etc., within 7 days prior to dosing or during the study
18. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes or known to prolong the QT interval
19. Consumption of products containing grapefruit within 10 days prior to dosing
20. Any special dietary changes during the 30 days prior to dosing, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor
21. Any strenuous exercise within 1 week of Check-in, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor
22. Known allergies to Na CMC or DMSO, components of the formulation to be used in this study
23. Current employment in a job requiring radiation-exposure monitoring
24. Participation in any study involving radioactivity within the last 12 months
25. More than one X-ray greater than the equivalent of one routine chest X-ray or one routine dental X-ray in the past 12 months
26. Donation of whole blood within 56 days prior to dosing
27. Plasma donation within 7 days prior to dosing
28. Participation in another clinical trial within 30 days prior to dosing
29. Hemoglobin < 12.0 g/dL
30. Previous use of PA-824

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Characterize the plasma pharmacokinetic variable area under the curve of a single oral-suspension dose of PA-824. | Days 0-12
  Characterize the plasma pharmacokinetics of a single oral-suspension dose of PA-824 in healthy adult male subjects by calculating the variable area under the curve [AUC (0-t)] from total PA-824 plasma concentrations.
Characterize the plasma pharmacokinetic variable maximum concentration of a single oral-suspension dose of PA-824. | Days 0-12
  Characterize the plasma pharmacokinetics of a single oral-suspension dose of PA-824 in healthy adult male subjects by calculating the variable maximum plasma concentration (Cmax) from total PA-824 plasma concentrations.
Characterize the plasma pharmacokinetic variable time to peak plasma concentration of a single oral-suspension dose of PA-824. | Days 0-12
  Characterize the plasma pharmacokinetics of a single oral-suspension dose of PA-824 in healthy adult male subjects by calculating the variable time to peak plasma concentration (Tmax) from total PA-824 plasma concentrations.

SECONDARY OUTCOMES:
The frequency and severity of treatment related adverse events throughout the study. | Days 0 -12
  In order to evaluate the safety and tolerability of a single oral-suspension dose of PA-824 in healthy adult male subjects

CONTACTS AND LOCATIONS:
Overall Officials: William Bridson, MD, Principal Investigator — Covance CRU
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States